CLINICAL TRIAL: NCT00530985
Title: Preserving Function Among Disability Applicants: A Motivational Enhancement Approach to Benefits Counseling
Brief Title: Preserving Function Among Disability Applicants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Rosen, Marc - Principal Investigator, Department of Veterans Affairs
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MR0024; MIRECC
Record Dates: First submitted 2007-09-16; First posted 2007-09-18 (Estimated); Last update posted 2009-07-02 (Estimated); Status verified 2009-06

CONDITIONS: Disability
Keywords: disability; substance abuse; vocational rehabilitation; case management
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Benefits Counseling
  Interventions: Behavioral: Benefits Counseling
- 2 (Active Comparator): VA Orientation
  Interventions: Behavioral: VA Orientation

INTERVENTIONS:
Behavioral: Benefits Counseling — Help deciding whether to work
  Arms: 1
Behavioral: VA Orientation — Orientation to services available at VA
  Arms: 2

SUMMARY:
To test the hypothesis that veterans counseled around managing their benefits will work more and have a better quality of life than those receiving non-specific counseling.

DETAILED DESCRIPTION:
The aim is to develop and test the efficacy of Benefits Counseling to improve quality of life among veterans who apply for VA benefits. Benefits Counseling involves providing claimants information about rehabilitation and work-related activities, benefits determination and management, and available substance abuse treatment . Benefits Counseling is designed to increase motivation to be active and promote engagement in substance abuse treatment. After enrolling 15 participants in an open-label pilot phase, 300 veterans who are not receiving benefits and are applying to VBA for disability benefits will be randomly assigned to Benefits Counseling or the control condition, VA Orientation, and both groups will be followed for one year.

The primary outcome measures will be observer-rated and self-rated quality of life. Secondary outcome measures will include substance use and treatment utilization.

ELIGIBILITY:
Inclusion Criteria:

1. Applying for VA service connection and not currently receiving VBA benefits.
2. Veterans who have been rated 0% service-connected but do not receive financial benefits are eligible to participate.
3. Able to provide valid consent
4. Age 18-65
5. Expresses willingness to discuss benefits with a counselor
6. Anticipates difficulty working

Exclusion Criteria:

1. Already receiving VA payments
2. Already receiving SSI or SSDI
3. Has a conservator

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2007-02; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Days engaged in work and work-related activities | 6 months

SECONDARY OUTCOMES:
substance use (as measured by days having used illicit drugs, alcohol to intoxication in the preceding days) | 6 months
treatment utilization (days in last 30 having participated in rehabilitation and work-related activities, number of days having participated in non-inpatient substance abuse treatment, number of days on any inpatient unit) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Marc I. Rosen, MD, Principal Investigator — VA Connecticut Health Care System (West Haven)
Locations (1):
- VA Connecticut Health Care System (West Haven), West Haven, Connecticut, United States